CLINICAL TRIAL: NCT05845515
Title: Laparoscopic Versus Open Orchiopexy in High Inguinal Undescended Testis, Prospective Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa AbdelRazek, Assistant Professor of Urology, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SVU/MED/URO016/1.21.4.184
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: We Conducted This Prospective Randomized Comparative Study to Compare Between Outcome of Laparoscopic and Open Orchiopexy of High Inguina
Keywords: laparoscopy , open , orchiopexy
MeSH Terms: interventions — Orchiopexy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic orchiopexy (Active Comparator): laparoscopic orchiopexy group
  Interventions: Procedure: laparoscopic orchiopexy
- open orchiopexy (Active Comparator): open orchiopexy group
  Interventions: Procedure: laparoscopic orchiopexy

INTERVENTIONS:
Procedure: laparoscopic orchiopexy — laparoscopic or open orchiopexy and comparison between the two groups

SUMMARY:
We conducted this prospective randomized comparative study to compare between outcome of laparoscopic and open orchiopexy of high inguinal.

All children presented to us with high inguinal undescended testis diagnosed by history, clinical examination and inguino-scrotal ultrasound were included in this study.

We exclude children with previous history of inguinal surgery or unfit for anesthesia.

150 patients with inclusion criteria were randomized (using block randomization method by Stata, version 13.1, StataCorp, for Microsoft Windows R) into two groups: Group A: 75 cases who were operated with laparoscopic orchiopexy. Group B: 75 cases who were operated with open orchiopexy.

All of the patients were subjected to the following: Complete history taking, and Clinical examination: High inguinal undescended testis, is testicle felt at upper half of inguinal canal and can't manipulated to the scrotum Pre-operative routine Laboratory investigation and Pre-operative imaging: Inguino-scrotal & colored Doppler ultrasound, were done for all patients. Patients were kept on fasting for 6 hours for solid food 2 hours for fluids before surgery. Informed written consent from all parents was obtained. All patients in our study underwent general anesthesia.

DETAILED DESCRIPTION:
Cryptorchidism, or undescended testis, is a common congenital anomaly in male child, it accounts 1 to 4.6% of full-term infants at the age of 1 year.

This condition usually involves the testicle that fail to travel from the abdomen through the inguinal canal to the scrotum during fetal life., cryptorchidism usually classified as inguinal cryptorchidism and intra-abdominal cryptorchidism in clinical practice, about 80% of undescended testis can feel the testis in the inguinal canal (1).

Cryptorchidism more than 6 months needs orchiopexy. Although laparoscopy has used widely in management of intra-abdominal cryptorchidism, there were controversy for its use in the treatment of inguinal cryptorchidism (1).

Open surgical treatment of such high inguinal testes is the most popular approach among urologists. Due to the difficult surgical mobilization of some high inguinal testes, as well as significant complications, including testicular retraction/atrophy (3-18%), we hypothesized in this study that laparoscopic orchiopexy for such high inguinal testes will be an attractive alternative approach (2).

Patients and methods

We conducted this prospective randomized comparative study to compare between outcome of laparoscopic and open orchiopexy of high inguinal.

All children presented to us with high inguinal undescended testis diagnosed by history, clinical examination and inguino-scrotal ultrasound were included in this study.

We exclude children with previous history of inguinal surgery or unfit for anesthesia.

150 patients with inclusion criteria were randomized (using block randomization method by Stata, version 13.1, StataCorp, for Microsoft Windows R) into two groups: Group A: 75 cases who were operated with laparoscopic orchiopexy. Group B: 75 cases who were operated with open orchiopexy.

All of the patients were subjected to the following: Complete history taking, and Clinical examination: High inguinal undescended testis, is testicle felt at upper half of inguinal canal and can't manipulated to the scrotum Pre-operative routine Laboratory investigation and Pre-operative imaging: Inguino-scrotal & colored Doppler ultrasound, were done for all patients. Patients were kept on fasting for 6 hours for solid food 2 hours for fluids before surgery. Informed written consent from all parents was obtained. All patients in our study underwent general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all children presented with high inguinal undescended testis

Exclusion Criteria:

* previous inguinal surgery
* unfit patients

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
success of laparoscopy and open surgery in treatment of high inguinal testis | 5 years
  assess the outcome and success rate of laparoscopy and open surgery in treatment of high inguinal testis

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No